CLINICAL TRIAL: NCT02834299
Title: A Randomized Controlled Study of a Dialectical Behavior Therapy Guided Self-Help Intervention for Binge Eating Disorder
Brief Title: Dialectical Behavior Therapy Guided Self-Help for Binge Eating Disorder
Acronym: DBT-GSH-BED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Jacqueline Carter-Major, Associate Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 3379
Record Dates: First submitted 2016-07-06; First posted 2016-07-15 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DBT Guided Self-Help (Experimental): Participants will be provided with the DBT self-help manual "Dialectical Behavior Therapy for Binge Eating: A Self-Help Program" by Safer, Adler & Masson (2016) and receive six brief therapy sessions via video-calling.
  Interventions: Behavioral: DBT Guided Self-Help
- DBT Unguided Self-Help (Experimental): Participants will be provided with the DBT self-help manual "Dialectical Behavior Therapy for Binge Eating: A Self-Help Program" by Safer, Adler & Masson (2016) and asked to follow the manual on their own.
  Interventions: Behavioral: DBT Unguided Self-Help
- Self-Esteem-Focused Unguided Self-Help (Active Comparator): Participants will be provided with the self-help manual "Self-Esteem" by McKay & Fanning (2016) as asked to follow the manual on their own.
  Interventions: Behavioral: Self-Esteem-Focused Unguided Self-Help

INTERVENTIONS:
Behavioral: DBT Guided Self-Help — DBT self-help manual plus six 30-minute therapy sessions for 12 weeks
  Arms: DBT Guided Self-Help
Behavioral: DBT Unguided Self-Help — DBT self-help manual without any therapy sessions for 12 weeks
  Arms: DBT Unguided Self-Help
Behavioral: Self-Esteem-Focused Unguided Self-Help — Self-esteem focused self-help manual without any therapy sessions for 12 weeks
  Arms: Self-Esteem-Focused Unguided Self-Help

SUMMARY:
This study will compare unguided and guided dialectical behavior therapy (DBT) self-help to an attention-placebo self-help control condition. Participants with binge eating disorder will be randomly assigned to one of the three self-help conditions for 12 weeks. Six guided self-help sessions will take place via secure video-calling. Assessments will take place before, mid-way through, and after the self-help program as well as at 3-month follow-up. Six guided self-help sessions will take place via secure video-calling.

DETAILED DESCRIPTION:
STUDY OBJECTIVES AND HYPOTHESES The primary objective of this randomized controlled trial is to compare the effectiveness of two methods of administering a dialectical behavior therapy (DBT) self-help intervention in a community sample of individuals with BED in NL: guided DBT self-help (DBT-GSH) and unguided DBT self-help (DBT-USH). A third condition designed to control for non-specific or common factors (e.g., receiving a self-help book) will also be included (NS-SH). This condition will be a self-help manual focused on improving low self-esteem using CBT strategies with no reference to binge eating.

METHODS

Sample size calculation:

Power analysis was based on the primary outcome variable: frequency of binge eating episodes. Assuming the three randomized groups (DBT-USH, DBT-GSH and NS-UGS) are equivalent at baseline, a between groups ANOVA will be used to compare them at post-treatment. Based on the findings of Masson et al. (2014), assuming an effect size of 0.40 and Type 1 error rate equal to .05, a sample size of at least 21 participants per group will yield 80% power. Assuming an attrition rate of 20%, we will require 25 participants per group.

Procedure:

Recruitment: Participants will be recruited from the community in the province of Newfoundland and Labrador (NL), Canada. Family doctor practices around the province will be informed about the study and brochures/posters will be sent to them. Posters advertising the study will be posted in hospitals, colleges, medical clinics, and universities. Advertisements will be placed on a local radio website and the PI will appear on the radio to advertise the study. Interested participants will be instructed to go to a website where they will fill in an initial screening questionnaire. Those who appear to meet the study inclusion criteria will be scheduled for an initial assessment interview via telephone or video-calling to confirm their eligibility.

Study inclusion/exclusion criteria:

Inclusion criteria: Participants will be male or female aged 18 and older who meet the DSM-5 diagnostic criteria for BED based on Eating Disorder Examination (Version 17). Additional inclusion criteria will include: 1) body mass index (BMI; kg/m2) of at least 18.5; 2) ability to read English; 3) high school graduate or equivalent; and 4) access to a computer, tablet or cell phone (with camera and microphone) and to high speed internet.

Exclusion criteria: Participants will be excluded for the following reasons: a) current specialized psychological treatment specifically for BED; b) current major medical illness that would interfere with treatment (e.g., cancer); c) current acute suicidal risk as assessed using the BDI-II ; d) current substance use disorder; and e) current psychotic symptoms . Individuals on a stable dose of antidepressant medication and/or sleep medication for at least 3 months will be eligible to take part.

Randomization: Participants will be randomized to one of the three intervention conditions (DBT-USH or DBT-GSH or NS-SH) using block randomization, with a block size of 5. Since no reliable predictors of BED outcome have been identified to date, we will not stratify the groups. The randomization list will be prepared by a research assistant not involved in the current study.

Interventions: Treatment will last 12 weeks in all conditions. Participants in both DBT self-help conditions will be provided with the DBT self-help manual "Dialectical Behavior Therapy for Binge Eating: A Self-Help Program". This manual is a self-help version of the well-established therapist-administered DBT treatment manual used in previous trials of DBT for BED. It consists of nine modules that aim to teach three skills to help participants stop binge eating: mindfulness, distress tolerance and emotion regulation. In the GSH condition, participants will receive six 30-minute one-on-one GSH sessions via a secure web-based video-calling program (Bluejeans) with a clinical psychology doctoral student therapist. GSH sessions will take place weekly for the first 2 weeks, biweekly for 6 weeks and then a final session will take place at week 12. The video-calling program allows GSH sessions to be recorded for supervision and treatment monitoring purposes. GSH therapists will have weekly group supervision meetings with the principal investigator to discuss any questions or challenges that arise. In both unguided self-help conditions, participants will be asked to do their best to follow the advice in the self-help manual on their own over the next 12 weeks.

Therapist Training and Supervision: After completing preparatory readings, therapists will attend a half-day training workshop with the principal investigator (JCM). Thereafter, therapists will meet weekly with JCM for group supervision to ensure competence and adherence to the GSH therapist manual.

Guided Self-Help (GSH) Therapist Manual. This manual was used in three previous CBT GSH trials, including one by the PI. It was adapted for the present study to guide therapists' DBT-GSH sessions.

Therapist Adherence to the GSH Therapist Manual: A random sample of 15% of video-taped GSH sessions will be reviewed by an independent rater to insure adherence to the Therapist Manual.

Participant drop-out: Consistent with an intention-to-treat approach, participants who drop out will be asked to continue to participate in the study assessments. To assess participant adherence, we will measure the number of times participants access the self-help manual website and the number of minutes they spend on each module. The number of eligible individuals who: decline to participate, are randomized, begin the study, or drop out of the study (and the week at which this occurs) will be recorded.

Assessment Measures: Except for the initial assessment interview, which will be conducted via video-calling, all study measures will be administered on-line via Qualtrics. Measures will be administered at baseline (Week 1), and post-treatment (Week12), as well as 3-month follow-up. A subset of measures (EDE-Q and DERS) will also be administered at mid-treatment (week 6).

Demographic variables:

Age, body weight, height, weight history, marital status, education level, ethnicity, age of onset of binge eating, and treatment history will be collected at baseline. Body weight will also be re-assessed at mid- and post-treatment.

Eating Disorder Psychopathology:

* Eating Disorder Examination Interview, Version 17 (EDE).
* Eating Disorder Examination Questionnaire (EDE-Q 6.0). General Psychological Distress
* Brief Symptom Inventory (BSI). Emotion Regulation
* Difficulties with Emotion Regulation Scale (DERS). Treatment Suitability and Expectancy (TSE)
* Perceived treatment suitability and expectations will be measured at baseline using two 10-point visual analogue scales used in previous self-help study on eating disorders.

Statistical analyses: The primary analysis will focus on the main outcome variable - number of binge eating episodes over the previous 28 days. If, after randomization, the three groups (i.e., GSH and USH) are equivalent at baseline, then an ANOVA will be used to compare the groups on binge eating frequency at post-treatment. Impact on eating disorder psychopathology, general psychological distress, quality of life, and difficulties with emotion regulation will also be examined. Eating disorder psychopathology, general psychological distress, quality of life, and difficulties with emotion regulation will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* meets DSM 5 criteria for binge eating disorder (BED)

Exclusion Criteria:

* receiving specialized psychological treatment for BED,
* BMI under 18.5,
* substance use disorder, major medical illness, psychotic symptoms

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire | Change from baseline at Week 12
  measures core eating disorder psychopathology and binge eating

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale | Change from baseline at Week 12
  Measures deficits in emotion management skills
Brief Symptom Inventory | Change from baseline at Week 12
  measures general psychological distress

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Carter, D.Phil., Principal Investigator — Memorial University
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: Undecided